CLINICAL TRIAL: NCT01349569
Title: Administration of an Allogeneic Myeloma GM-CSF Vaccine in Conjunction With a Lenalidomide Containing Regimen in Myeloma Patients With Near Complete Remission
Brief Title: Allogeneic GM-CSF Vaccine and Lenalidomide in Treating Myeloma Patients With Near Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1115; NA_00044463 (Other: JHMIRB)
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myeloma Vaccine, Prevnar, & Lenalidomide (Experimental): Lenalidomide will be continued on the same dose as was being administered prior to the study. The allogeneic myeloma vaccine and Prevnar-13 vaccine will be given on four days over the course of the study.
  Interventions: Drug: Lenalidomide; Biological: Allogeneic Myeloma Vaccine; Biological: Prevnar-13

INTERVENTIONS:
Drug: Lenalidomide — Dosage forms: 5, 10, 15 and 25 mg capsules. Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5- 25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Other Names: Revlimid
Biological: Allogeneic Myeloma Vaccine — A total of 4 vaccines will be administered. The first three at monthly intervals and a booster at 6 months from the initial vaccine. Each vaccination will consist of five total intra-dermal injections, two each in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). Each dose will be administered on an outpatient basis. The subject must be observed in the clinic for at least 30 minutes after vaccination is completed.
Biological: Prevnar-13 — Prevnar-13 will be administered at 0.5ml dose by intramuscular injection at the same time as GVAX vaccine.
  Other Names: Pneumococcal 13-Valent Conjugate Vaccine

SUMMARY:
This research is being done to find out if the investigators can improve outcomes for multiple myeloma patients by giving a myeloma vaccine to patients who are already on lenalidomide (Revlimid) and in a near complete remission.

DETAILED DESCRIPTION:
This is a single institution, single arm, Phase II study examining the clinical efficacy of an allogeneic GM-CSF secreting myeloma vaccine in combination with lenalidomide. Fifteen (15) patients enrolled in the study must have two disease measurements (including the last one) consistent with a near complete remission (M-spike negative with persistence of immunofixation) per criteria for response in a 6 month period. Patients will continue on the dose of lenalidomide they were on prior to being enrolled but will need to discontinue steroids for at least 4 weeks. Patients will receive 4 vaccinations on day 14(+/-3 days) of cycles 1, 2, 3 and 6 from enrollment that will include both the myeloma vaccine as well as Prevnar.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma eligibility criteria are the following:

  * sustained near complete remission (nCR) for 4 months defined as no measurable M-spike and a positive immunofixation
  * early biochemical relapse as manifest by going from a true CR (immunofixation negative) to a nCR (immunofixation positive) at any time
  * conversion from a nCR to the appearance of a monoclonal spike in the serum not greater than 0.3mg/dL
* age 18 years and older
* Eastern Cooperative Oncology Group performance scores 0-2
* History of measurable serum or urine M protein or free light chains
* Life expectancy greater than 12 months
* Corrected serum calcium < 11 mg/dL, and no evidence of symptomatic hypercalcemia
* Serum creatinine< 2
* Absolute Neutrophil Count >1000
* Platelet >100,000
* Total bilirubin less than or equal to 1.5 x Upper limit of normal
* Aspartate aminotransferase and Alanine transaminase less than or equal to 3 x Upper limit of normal
* Negative pregnancy test if applicable
* Ability to comprehend and have signed the informed consent.
* Disease free of prior malignancies for < 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to aspirin may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Disease progression after stopping corticosteroids as defined as the appearance of an M-spike >0.5g/dL
* Patients with a known diagnosis of POEMS syndrome, plasma cell leukemia, non-secretory myeloma and amyloidosis.
* HIV disease, active infection requiring treatment with antibiotics, anti-fungal or anti-viral agents within 2 weeks of enrollment would be excluded from the study.
* Patients who have participated in any clinical trial, within four weeks prior to registration on this trial, which involved an investigational drug.
* History of an active malignancy other than myeloma
* Autoimmune disease requiring active treatment.
* Known contra-indication to any component of Prevnar 13 including the diphtheria toxoid-containing vaccine.
* History of latex allergy
* History of an autologous stem cell transplant within the past 12 months or less
* History of an allogeneic transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borrello, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were screen failures. One participant withdrew consent prior to starting the study.
Groups:
- Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide: Lenalidomide: Dosage forms: 5, 10, 15 and 25 mg capsules. Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5- 25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Allogeneic Myeloma Vaccine: A total of 4 vaccines will be administered. The first three at monthly intervals and a booster at 6 months from the initial vaccine. Each vaccination will consist of five total intra-dermal injections, two each in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). Each dose will be administered on an outpatient basis. The subject must be observed in the clinic for at least 30 minutes after vaccination is completed.
  Prevnar-13: Prevnar-13 will be administered at 0.5ml dose by intramuscular injection at the same time as GVAX vaccine.
Period: Overall Study
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
Started | 16
Completed | 12
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Population: One participant withdrew consent prior to receiving the study intervention, leaving sixteen participants who received at least one day of intervention.
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 68 [45 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Response Conversion Rate
Description: Number of participants who converted from near complete remission (nCR) to complete remission (CR) as measured by the International Myeloma Working Group Uniform Response Criteria. Near complete remission is defined as negative serum and urine electrophoresis, < 5% plasma cells in the bone marrow, and positive serum and/or urine immunofixation. Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
Time Frame: Up to 1 year
Population: Out of the 16 baseline participants, one received only one dose of vaccine and then had progression of disease. He was replaced and not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
Number analyzed (Participants) | 15
Participants | 8

2. Secondary Outcome: Time to Response
Description: Median time for conversion of response from near complete remission (nCR) to complete remission (CR) as measured by the International Myeloma Working Group Uniform Response Criteria. Near complete remission is defined as negative serum and urine electrophoresis, < 5% plasma cells in the bone marrow, and positive serum and/or urine immunofixation. Complete response is defined as negative serum and urine immunofixation and a bone marrow aspirate with < 5% plasma cells.
  as measured by immunofixation converting from positive to negative.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
Number analyzed (Participants) | 15
months | 11.7 [2 to 47]

3. Secondary Outcome: Effect on Clonogenic Myeloma Precursors
Description: Measures of stem cell population and plasma cell population.
Time Frame: Baseline, Cycle 3 Day 14, Cycle 6 Day 14, and 1 year
Population: Data was not collected for this outcome measure due to technical difficulties in the assay.
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Grade 3-4 Toxicity
Description: Number of participants who experienced grade 3-4 toxicity as per CTCAE 4.0.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
Number analyzed (Participants) | 16
Participants | 0

5. Secondary Outcome: Tumor-specific Immunity as Assessed by Percentage of CD3+/CSFSE-low/IFN-gamma+ Cells
Description: Immunity is measured by the percentage of CD3+/CSFSE-low/IFN-gamma+ cells. A positive result for a given participant is defined as greater than two standard deviations above that participant's baseline. The data are presented as three groups because the responses were analyzed separately, but all participants were part of the single study arm as represented by the remainder of the record. GVAX-specific immune response and Prevnar-specific immune response was assessed in the same patient by using GVAX and Prevnar-specific co-markers.
Time Frame: Baseline, Cycle 3 Day 14, end of study (up to 1 year)
Population: Out of the 16 baseline participants, one received only one dose of vaccine and then had progression of disease. He was replaced and not included in this analysis. Only 8/15 participants experienced complete response (CR), therefore only 8 participants analyzed in the CR rows and 7 participants analyzed in the progressive disease (PD) rows.
Measure: Mean (Standard Deviation); unit: percentage of cells
Groups:
- Pre-vaccine (Baseline): Lenalidomide: Dosage forms: 5, 10, 15 and 25 mg capsules. Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5- 25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
- GVAX Vaccine: Allogeneic Myeloma Vaccine: A total of 4 doses will be administered. The first three at monthly intervals and a booster at 6 months from the initial dose. Each vaccination will consist of five total intra-dermal injections, two each in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). Each dose will be administered on an outpatient basis. The subject must be observed in the clinic for at least 30 minutes after vaccination is completed.
- Prevnar Vaccine: Prevnar-13 will be administered at 0.5ml dose by intramuscular injection at the same time as GVAX vaccine.
Arm/Group | Pre-vaccine (Baseline) | GVAX Vaccine | Prevnar Vaccine
Number analyzed (Participants) | 15 | 15 | 15
percentage of cells
  Complete Response (CR) patients at Baseline: number analyzed (Participants) | 8 | 8 | 8
  Complete Response (CR) patients at Baseline | 1.2 (0.4) | 0.36 (0.6) | 0 (NA) — Mean percentage of CD3+/CSFSE-low/IFN-gamma+ cells was zero, therefore no standard of deviation
  CR patients at Cycle 3 Day 14: number analyzed (Participants) | 8 | 8 | 8
  CR patients at Cycle 3 Day 14 | 7.3 (2.6) | 13.3 (3) | 4.54 (2.1)
  CR patients at end of Study: number analyzed (Participants) | 8 | 8 | 8
  CR patients at end of Study | 6.3 (1.4) | 13.7 (5.1) | 3.6 (1.4)
  Progressive Disease (PD) patients at Baseline: number analyzed (Participants) | 7 | 7 | 7
  Progressive Disease (PD) patients at Baseline | 0.43 (0.44) | 0.45 (0.7) | 0 (NA) — Mean percentage of CD3+/CSFSE-low/IFN-gamma+ cells was zero, therefore no standard of deviation
  PD patients at Cycle 3 Day 14: number analyzed (Participants) | 7 | 7 | 7
  PD patients at Cycle 3 Day 14 | 1.7 (2.9) | 5.7 (1.4) | 0 (NA) — Mean percentage of CD3+/CSFSE-low/IFN-gamma+ cells was zero, therefore no standard of deviation
  PD patients at end of study: number analyzed (Participants) | 7 | 7 | 7
  PD patients at end of study | 0.4 (0) | 0.21 (0) | 1.7 (0)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse events were assessed every 28 days.
Groups:
- Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide: Lenalidomide: Dosage forms: 5, 10, 15 and 25 mg capsules. Patients will be continued on the same dose of lenalidomide as they were prior to being enrolled in the study. Doses of lenalidomide for investigation can vary from 5- 25 mg/day, orally on days 1 - 21 followed by 7 days rest (28 day cycle).
  Allogeneic Myeloma Vaccine: A total of 4 vaccines will be administered. The first three at monthly intervals and a booster at 6 months from the initial vaccine. Each vaccination will consist of five total intra-dermal injections, two each in the right and left anterior upper thighs, and one in the non-dominant upper arm (unless contraindicated). Each dose will be administered on an outpatient basis. The subject must be observed in the clinic for at least 30 minutes after vaccination is completed.
  Prevnar-13 will be administered at 0.5ml dose by intramuscular injection at the same time as GVAX vaccine.
Arm/Group | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide (N=16)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloma Vaccine, Prevnar-13 Vaccine, & Lenalidomide (N=16)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pressure (Cardiac disorders) | 1 (1)
Pain - chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Peripheral edema (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 3 (3)
Injection site reactions (Skin and subcutaneous tissue disorders) | 15 (40)
Interface haze (Eye disorders) | 1 (1)
Lump - left wrist (Skin and subcutaneous tissue disorders) | 1 (1)
Cramping (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain - knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - mouth (Gastrointestinal disorders) | 1 (1)
Pain - right side (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3)
Pain - abdomen (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes